CLINICAL TRIAL: NCT06379490
Title: Effect of Ultrasound-guided Lateral Infraclavicular Brachial Plexus Block With Lidocaine or Ropivacaine for Closed Reduction of Distal Radius Fractures - A Randomized Controlled Non-inferiority Trial
Brief Title: Ultrasound-guided Infraclavicular Block With Lidocaine or Ropivacaine for Closed Reduction of Distal Radius Fractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTA no: 2024-510572-20-00; 2024-510572-20-00 (EU CTIS Number); P-2023-296 (Other: Privacy - Region Hovedstaden)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Distal Radius Fractures; Lidocaine; Ropivacaine; Fracture Dislocation; Closed Reduction of Fracture and Application of Plaster Cast; Colles' Fracture
Keywords: anesthetics, local; regional anesthesia; peripheral nerve block; brachial plexus block; lateral infraclavicular block; closed reduction; distal radius fracture; colles' fracture; wrist fracture
MeSH Terms: conditions — Wrist Fractures; Fracture Dislocation; Colles' Fracture | interventions — Ropivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ropivacaine 5 mg/ml (Active Comparator): 30 ml of ropivacaine 5 mg/ml (Injectable solution - perineural administration - only once)
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- Ropivacaine 2 mg/ml (Experimental): 30 ml of ropivacaine 2 mg/ml (Injectable solution - perineural administration - only once)
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Lidocaine 10 mg/ml (Experimental): 30 ml of lidocaine 10 mg/ml with epinephrine 5 μg/ml (Injectable solution - perineural administration - only once)
  Interventions: Drug: Lidocaine epinephrine

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — 30 ml of Ropivacaine 0.2% = 60 mg ropivacaine
  Other Names: Ropivacaine 2 mg/ml
  Arms: Ropivacaine 2 mg/ml
Drug: Lidocaine epinephrine — 30 ml of Lidocaine 1% with 5 μg/ml epinephrine = 300 mg lidocaine + 150 μg epinephrine
  Other Names: Lidocaine 10 mg/ml
  Arms: Lidocaine 10 mg/ml
Drug: Ropivacaine 0.5% Injectable Solution — 30 mL of Ropivacaine 0.5% = 150 mg Ropivacaine
  Other Names: Ropivacaine 5 mg/ml
  Arms: Ropivacaine 5 mg/ml

SUMMARY:
To investigate the feasibility of the lateral infraclavicular plexus brachialis (LIC) block for acute closed reduction of distal radius fractures, the investigators will compare the pain-relieving and muscle-relaxing properties of the LIC block with short- and long-acting local anesthetics in different concentrations but at the same volume. In addition to motor and sensory blockade during repositioning, feasibility will also be assessed by other patient-related and block-related factors, as well as by factors related to the repositioning and plastering procedure.

ELIGIBILITY:
Inclusion Criteria:

Patients who have given written informed consent to participate in the study after having understood it, as well as:

• Having a distal radius fracture requiring closed reduction

Exclusion Criteria:

Patients who meet one or more of the following criteria will be excluded from participating in the study:

* BMI > 40 kg/m2
* Weight < 50 kg
* Age < 18 years
* American Society of Anesthesiologists (ASA) physical status classification system grade >3
* Allergy to experimental drugs
* Patients who cannot cooperate with the examinations or treatment
* Patients who do not understand or speak Danish
* Patients with peripheral or central neurological disease or nerve damage with neurological effect on the upper extremity, where closed reduction is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Block success | 45 minutes after block performance
  The incidence of successful blockade 45 minutes after block performance.
  The following 4 nerves will be tested: radial, musculocutaneous, ulnar and median nerves.
  Sensory blockade assessment:
  * A 3-point scale is used for cold sensation assessment: 1 point = normal sensation of cold, 2 points = reduced sensation of cold and 3 points = no cold sensation.
  * A complete sensory blockade is defined as all four nerves obtaining 3 points (no cold sensation).
  Motor blockade assessment:
  * Assessment is done using a 4-point Manual Muscle Testing Scale: 3 points = no difference, the movement against resistance is possible, 2 points = a slight difference, the movement against slight resistance is possible, 1 point = movement is significantly compromised, 0 points = paralysis.
  * A complete motor blockade is defined as all four nerves obtaining: 1 point or 0 points.
  Successful blockade:
  • Complete sensory and motor blockade 45 minutes after block performance.

OTHER OUTCOMES:
Degree of sensory and motor blockade | 30 to 45 minutes after block performance
  Degree of sensory and motor blockade 30 and 45 minutes after block performance.
  Sensory blockade assessment:
  * A 3-point scale is used for cold sensation assessment: 1 point = normal sensation of cold, 2 points = reduced sensation of cold and 3 points = no cold sensation.
  * A complete sensory blockade is defined as all four nerves obtaining 3 points (no cold sensation).
  Motor blockade assessment:
  * Assessment is done using a 4-point Manual Muscle Testing Scale: 3 points = no difference, movement against resistance is possible, 2 points = a slight difference, movement against slight resistance is possible, 1 point = movement is significantly compromised, 0 point = paralysis.
  * A complete motor blockade is defined as all four nerves obtaining: 1 point or 0 points.
Total duration of sensory blockade | 24 hours after completed block performance
  From the completion of the LIC block until the ending of the sensory blockade.
  Duration in hours:minutes.
Total duration of motor blockade | 24 hours after completed block performance
  From the completion of the LIC block until the ending of motor blockade.
  Duration in hours:minutes.
Pain intensity before block performance | Up to 45 minutes after inclusion interview
  Pain intensity measured before block performance with a numeric rating scale (NRS 0 - 10 (0 = no pain; 10 = worst pain imaginable))
Time to pain relief/lowest pain intensity | Up to 45 minutes after block performance
  Time to pain relief/lowest pain intensity after block performance and before performing the closed reduction
  Duration in hours:minutes
Pain intensity during closed reduction | Duration of closed reduction (approx. 5 to 10 minutes)
  Pain intensity measured during closed reduction with a numeric rating scale (NRS 0 - 10 (0 = no pain; 10 = worst pain imaginable))
Pain intensity during cast application | Duration of cast application (approx. 5 to 10 minutes)
  Pain intensity measured during cast application with a numeric rating scale (NRS 0 - 10 (0 = no pain; 10 = worst pain imaginable))
Time to pain breakthrough after the blockade has ended | Up to 24 hours after block performance
  Time after block performance until pain breakthrough defined as NRS>3 (NRS 0 - 10 (0 = no pain; 10 = worst pain imaginable))
  Duration in hours:minutes
Maximum pain intensity after the blockade has ended | Up to 24 hours after block performance
  Pain intensity measured after the blockade has ended with a numeric rating scale (NRS 0 - 10 (0 = no pain; 10 = worst pain imaginable))
Duration of maximum pain intensity after the blockade has ended | Up to 24 hours after block performance
  Time period of maximum pain intensity after the blockade has ended
  Duration in hours:minutes
Amount of strong painkillers consumed by patients within 24 hours after closed reduction | 24 hours after completed block performance
  Amount of strong painkillers consumed by patients within 24 hours after closed reduction will be measured in 24-hour morphine equivalents (milligrams).
Grading of closed reduction difficulty | Duration of closed reduction (approx. 5 to 10 minutes)
  Grading of closed reduction difficulty measured with a numeric rating scale (NRS 0 - 10 (0 = no difficulty; 10 = very difficult))
Quality of closed reduction evaluated by X-ray imaging | 24 hours and 30 days after block performance
  Quality of closed reduction evaluated by X-ray imaging using the following radiological criteria:
  * More than 10 degrees of dorsal angulation of the articular surface of the radial in a side view as compared to perpendicular to the longitudinal axis of the radial
  * Ulnar variance of more than 2 mm
  * Articular step-off of more than 2 mm
  * Incongruity of the distal radioulnar joint
  * Loss of substance/comminuted fracture of the dorsal cortex
Attempts used for closed reduction | Up to 4 hours after block application
  Number of attempts used for closed reduction. One attempt is defined as closed reduction before X-ray control imaging.
Grading of casting difficulty | Duration of cast application (approx. 5 to 10 minutes
  Grading of casting difficulty measured with a numeric rating scale (NRS 0 - 10 (0 = no difficulty; 10 = very difficult))
The patient's experience of the treatment | Up to 24 hours after block performance
  The patient's experience of the treatment using a numeric rating scale (NRS 0 - 10 (0 = very dissatisfied; 10 = very satisfied))
Occurence of adverse events (AE) and serious adverse events (SAE) | 24 hours and 30 days after block performance
  Adverse events are defined as any harmful or unwanted events, signs, or symptoms that occur during participation in the study period.
  Serious adverse events are defined as events resulting in death, a life-threatening condition, permanent disability, hospital admission, or prolonged hospital admission.
  Based on phone interviews and medical records 24 hours and 30 days after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anders K. Nørskov, PhD, Principal Investigator — Copenhagen University Hospital - North Zealand
Locations (1):
- Copenhagen University Hospital - North Zealand, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No